CLINICAL TRIAL: NCT03614650
Title: Antigen-specific Engineered Immune Effector Cells (EIE) Against Gastro-Intestinal (GI) Cancer
Brief Title: Immunotherapy Treating GI Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-18002
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: immunotherapyT cellGI cancergene therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIE cells to treat cancer (Experimental): EIE cells to treat cancer
  Interventions: Biological: engineered immune cells

INTERVENTIONS:
Biological: engineered immune cells — Engineered immune effector cells (EIE)

SUMMARY:
The primary objectives are to evaluate the safety and efficacy of infusion of autologous gastro-intestinal (GI) cancer antigen-specific engineered immune effector cells (EIE).

DETAILED DESCRIPTION:
Gastro-intestinal (GI) cancer is becoming the top-ranked high mortality cancer in recent years. Every year, approximate 5,300,000 people in China are diagnosed with cancer, of which about 2,000,000 die each year, and esophagus cancer, gastric cancer and colorectal cancer account for ~50% of all GI cancer cases. GI cancer causes 500 thousand deaths a year. In China, nearly 85% of patients with cancer of the digestive tract are in middle to late stage at diagnosis. Regardless of the treatment, the five year survival rate is only 36%. GI cancers include cancer in the oral cavity, pharynx, esophagus, stomach, small intestine (duodenum, jejunum, ileum) and large intestine (cecum, colon, rectum). The main malignant tumors of the GI tract are esophageal, gastric, colorectal, liver, and pancreatic cancer.

Adoptive immunotherapy based on cytotoxic T lymphocytes reactive with specific antigens has proven to be effective in many studies. In vitro induction of cancer antigen-specific immune cells and genetic engineering of target specific immune cells have great potential for cancer eradication. This study aims to evaluate the safety and efficacy of ex vivo manipulated EIE cells including chimeric antigen receptor (CAR) modified immune cells in treating cancer. The primary study objectives are to evaluate the safety of the investigational product, autologous EIE cells, to subjects by intravenous and intratumoral injections. The secondary study objectives are (1) to evaluate the success rate of generating autologous EIE cells ex vivo, and (2) to determine the anti-cancer efficacy of the EIE cells.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written, informed consent obtained prior to any study-specific procedures. 2. The results of immune staining of the patient's cancer specimens positive for any one or more of tumor-associated antigens, such as GD2, mesothelin, CEA, P16, MMP, Melan A, MAGE A1, MAGE A3, and MAGE A4.

  3. Eastern Cooperative Oncology Group (ECOG) PS of 0, 1 or 2. 4. Life expectancy ≥ 3 months. 5. Able to comply with the protocol. 6. Histologically confirmed and documented high risk International Federation of Gynecology and Obstetrics (FIGO): Stage III-IV.

  7. Not pregnant, and on appropriate birth control if of childbearing potential. 8. Adequate bone marrow reserve with

  • absolute neutrophil count (ANC) ≥ 1000/mm3.• Platelets ≥100,000/mm3. 9. Adequate renal and hepatic function with• Serum creatinine ≤ 2 x upper limit of normal (ULN).• Serum bilirubin ≤ 2 x ULN.• aspartate aminotransferase (AST)/ALT ≤ 2 x ULN.• Alkaline phosphatase ≤ 5 x ULN.• Serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.

Exclusion Criteria:

* 1. The results of immune staining of the patient's tumor-associated antigens are all negative.

  2. Participation in any other cell therapy protocols within one year. 3. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug.

  4. Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).

  5. Pregnant or lactating females. 6. Unable to comply with the trial related requirement. 7. Inadequate bone marrow function:
  * Absolute neutrophil count < 1.0 x 10e9/L.
  * Platelet count < 100 x 10e9/L.
  * Hb < 9 g/dL.

Inadequate liver and renal function:

* Serum (total) bilirubin > 1.5 x ULN.• AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases).
* Alkaline phosphatase > 2.5 x ULN (or > 5 x ULN in case of liver metastases or > 10 x ULN in case of bone metastases).
* Serum creatinine >2.0 mg/dl (> 177 μmol/L).
* Urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.

  8. Serious active infection requiring i.v. antibiotics during screening. 10. Subject infected with HIV (HIV antibody positive), Treponema pallidum antibody positive or TB culture positive.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of adverse effects after EIE cell injection | up to one month
  To assess the safety of autologous EIE cells in patients. The percentage of patients who have adverse effects will be evaluated by using the NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Rate of successful EIE generation | up to one month
  The percentage of successful EIE generation, which are derived from subjects and pass the safety test after standard culture procedures, viable for at least one preparation, will be evaluated.
Ability of EIE cells to reduce cancer burden | after 1 month from EIE cells infusion until 12 months after infusion
  measurement of tumor marker in blood and examination of tumor size change
The anti-cancer effects | after 1 month from EIE cells infusion until 24 months after infusion
  Objective response (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. CR is disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Study Chair — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No